CLINICAL TRIAL: NCT05055063
Title: A Phase 1 With Extension Cohort, Single Arm, Single Center, Open Label Trial of Belantamab Mafodotin for the Treatment of High-Risk Smoldering Multiple Myeloma (BELLA)
Brief Title: A Phase 1 With Extension Cohort, Single Arm, Single Center, Open Label Trial of Belantamab Mafodotin for the Treatment of High-Risk Smoldering Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0431; NCI-2021-08991 (Other: NCI-CTRP Registry Program)
Record Dates: First submitted 2021-09-07; First posted 2021-09-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin (Experimental): belantamab mafodotin by vein over 30-60 minutes on Day 1 of each 56-day cycle for the first 6 cycles.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — by vein over 30-60 minutes on Day 1 of each 56-day cycle for the first 6 cycles.

SUMMARY:
This is a single-center, single arm, phase I study designed to determine the safety and find the recommended Phase 2 dose (RP2D) or maximum dose level (MTD) of Belantamab Mafodotin in patients with high-risk smoldering multiple myeloma. The study will have a dose-finding part and a dose-expansion part. The maximum number of enrolled patients will be 30 with 18 patients for the dose-finding part and 12 patients for the dose-expansion part. Once we determine the MTD or RP2D in the dose-finding part, we will enroll and treat 12 additional patients at the MTD or RP2D in the expansion part. Efficacy will be assessed through the overall response rate (ORR) at the end of the study. With the limited number of patients for the dose-expansion part, we will not have formal futility monitoring rule.

DETAILED DESCRIPTION:
Primary Objective: To obtain the recommended Phase 2 dose (RP2D) or maximum tolerated dose of single agent belantamab mafodotin in high risk SMM.

Secondary Objectives: Overall response rate per International Myeloma Working Group (IMWG) criteria. Progression free survival at 2 years, overall survival, duration of response, safety and clinical benefit rate.

Exploratory Studies: Evaluate correlative endpoints including immune, cellular and molecular profiling, minimal residual disease, BCMA staining of bone marrow, pharmacokinetics, pharmacodynamics and mechanisms of resistance to belantamab mafodotin.

ELIGIBILITY:
Inclusion Criteria:

Patients must be diagnosed with high-risk smoldering multiple myeloma (SMM) as confirmed by the following (all three must be present):

1. Bone marrow plasmacytosis with ≥ 10% plasma cells in bone marrow biopsy
2. Immunoparesis (reduction in at least one uninvolved immunoglobulin in blood)
3. ≥ 95% aberrant plasma cells of all plasma cells by flow cytometry of the bone marrow aspirate

   * Creatinine clearance (CrCl) ≥ 30 ml/min. CrCl will be calculated using the Modification of Diet in Renal Disease (MDRD) equation.
   * Age ≥ 18 years.
   * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
   * Absolute neutrophil count (ANC) ≥ 1.0 x 109 /L, hemoglobin more or equal than 2 grams below the institutional level of normal and platelet count ≥ 90 x 109/L. Platelet and blood transfusions are allowed on protocol. Growth factors, including granulocyte colony stimulating factors and erythropoietin are allowed.
   * Adequate hepatic function, with bilirubin ≤ 1.5 x the ULN, and AST and ALT ≤ 2.5 x ULN.
   * Females of childbearing potential are eligible to participate if they agree to avoid pregnancy by using an adequate method of contraception that is highly effective with a failure rate of <1% per year (2 barrier method or 1 barrier method with a spermicide or intrauterine device during and for 4 months after the last dose of belantamab mafodotin). Adequate methods of contraception are provided as examples. Other acceptable and effective methods of birth control are also permitted (eg, abstinence). Women of child bearing potential must have a negative serum pregnancy test result within 72 hours prior to the first administration of belantamab mafodotin and at the end of treatment visit. A negative urine pregnancy test is required prior to each subsequent belantamab mafodotin dose administration
   * Females of childbearing potential are eligible to participate if they agree to notdonate eggs (ova, oocytes) for the purpose of reproduction during the study and for 4 months after the last dose of belantamab mafodotin.
   * Male participants are eligible to participate if they agree to the following from the time of first dose of belantamab mafodotin until 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

     * be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent,
     * OR must agree to use contraception/barrier as follows:
     * agree to use a male condom, even if they have undergone a successful vasectomy
     * and female partner of childbearing potential to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse.
   * Men must agree to not donate sperm while on the study and for at least 6 months after the last dose of belantamab mafodotin.
   * Subjects must be able to give informed consent.
   * Subjects must be either newly diagnosed smoldering myeloma or not have received prior or concurrent treatment for smoldering multiple myeloma with chemotherapy agents approved for the treatment of smoldering multiple myeloma. Patients who have been treated previously on a clinical trial or with non-approved agents for their smoldering myeloma can be included.
   * Exclusion Criteria:
   * Evidence of myeloma defining events or biomarkers of malignancy due to underlying plasma cell proliferative disorder meeting at least one of the following:

     * Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
     * Renal Insufficiency: creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL
     * Anemia: hemoglobin value more than 2 g/dL < normal reference
     * Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT).
     * Clonal bone marrow plasma cell percentage ≥ 60%
     * Involved: uninvolved serum free light chain ratio ≥100 measured by Freelite assay (The Binding Site Group, Birmingham, UK)
     * >1 focal lesions on MRI studies (each focal lesion must be 5 mm or more in size)
   * Bisphosphonates are permitted, including pamidronate, zoledronic acid, alendronate, ibandronate, risedronate.
   * Treatment with corticosteroids is not permitted, unless the patient is on a stable chronic dose of inhaled steroids to treat respiratory diseases or on stable chronic steroid replacement therapy for endocrinology disorders. Steroids may be used treat infusion related reactions. Inhaled, intranasal, and topical ophthalmic steroids are not prohibited.
   * Radiotherapy is not permitted.
   * Prior or concurrent treatment for smoldering multiple myeloma with chemotherapy agents approved for the treatment of smoldering multiple myeloma
   * Plasma cell leukemia
   * Pregnant or lactating females. It is not known whether belantamab mafodotin is excreted in human milk. The effect of belantamab mafodotin of newborns/infants is unknown. Women should be advised to discontinue breast-feeding prior to initiating treatment with belantamab mafodotin and for at least 70 days after the last dose. These potential risks may also apply to other agents used in this study.
   * Active hepatitis B or C infection
   * Known HIV infection
   * Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin
   * Concurrent treatment with other anti-cancer therapy is not permitted
   * Has significant cardiovascular disease with:

     * NYHA Class III or IV symptoms,
     * uncontrolled hypertension
     * hypertrophic cardiomyopathy restrictive cardiomyopathy, or myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months prior to enrollment
     * evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block as determined by history and physical examination.
   * Uncontrolled intercurrent illness including but not limited to active infection requiring treatment or psychiatric illness/social situations that would compromise compliance with study requirements
   * Contraindication to any concomitant medication, including pre-medications or hydration given prior to therapy
   * Major surgery within 1 month prior to enrollment
   * Previous or concurrent malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
   * Presence of active renal condition (infection, requirement for dialysis, or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting are eligible, provided they fulfil renal criteria provided above.
   * Any evidence of active mucosal or internal bleeding
   * Received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of belantamab mafodotin
   * Cirrhosis or current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
   * Current corneal epithelial disease except mild changes in corneal epithelium
   * Use of contact lenses while participating in this study, except at the direction of the study MD/OD
   * Severe dry eye patients and monocular patients are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To establish the recommended Phase 2 dose (RP2D) or maximum tolerated dose of single agent belantamab mafodotin in high risk SMM. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org